CLINICAL TRIAL: NCT04331587
Title: Evaluation of Thin and Ultrathin Bronchoscopy With Transbronchial Needle Aspiration and Radial Probe Endobronchial Ultrasound for Peripheral Pulmonary Lesions
Brief Title: Thin and Ultrathin Bronchoscopy With Transbronchial Needle Aspiration and Radial Probe Endobronchial Ultrasound for Peripheral Pulmonary Lesions
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Olympus (Industry)
Responsible Party: Sponsor
Other Study IDs: 202003071
Record Dates: First submitted 2020-03-27; First posted 2020-04-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Peripheral Pulmonary Nodules

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Bronchoscopy: The bronchoscopy procedure and use of both the thin and ultrathin bronchoscopes are considered standard of care and will be performed under moderate sedation in an outpatient bronchoscopy suite as part of each patient's clinical care.
  Interventions: Device: BF-P190 4 mm thin bronchoscope; Device: BF-MP190F 3 mm ultrathin bronchoscope; Device: Radial ultrasound probe (UM S20-17S); Device: PeriView FLEX 21G Single Use Aspiration Needle

INTERVENTIONS:
Device: BF-P190 4 mm thin bronchoscope — * EVIS EXERA III Bronchofiberviedoscopes
  * Olympus
Device: BF-MP190F 3 mm ultrathin bronchoscope — * EVIS EXERA III Bronchofiberviedoscopes
  * Olympus
Device: Radial ultrasound probe (UM S20-17S) — -Olympus
Device: PeriView FLEX 21G Single Use Aspiration Needle — * NA-403D-2021
  * Gyrus ACMI, Inc.

SUMMARY:
To collect data on diagnostic yield of thin and ultrathin bronchoscopes with radial probe endobronchial ultrasound (radial EBUS) and transbronchial needle aspiration (TBNA) during routine standard of care bronchoscopy for peripheral pulmonary lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 and older
* Patients presenting with peripheral pulmonary lesions 1-7cm in greatest diameter on axial CT or PET scan in need of bronchoscopic biopsy for clinical purposes

Exclusion Criteria:

* Patients who are unable to undergo flexible bronchoscopy as determined by the bronchoscopist prior to the procedure
* Patients unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being seen at Washington University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
Overall diagnostic yield (concentric and eccentric lesions) for peripheral pulmonary nodules | Receipt of cytology/histopathology results (approximately 7 days)
  -To determine overall diagnostic yield (concentric and eccentric lesions) for peripheral pulmonary nodules utilizing using a standard of care combined approach of 4mm thin and 3mm ultrathin bronchoscopes with TBNA and radial EBUS and compare it to a historical baseline diagnostic yield of 60% established at Washington University School of Medicine (WUSM) when using TBNA and radial EBUS and a 4mm thin bronchoscope.

SECONDARY OUTCOMES:
Incidence of related adverse events | Up to 4 days following procedure
  -Adverse events related to the bronchoscopy procedure and/or devices used during the procedure (bronchoscope, radial EBUS, PeriView Flex needle).
Procedure time measured in minutes from oral scope insertion to scope removal upon completion of the bronchoscopy procedure | From start of procedure through end of procedure (day 1)
Size of target lesions measured at the greatest diameter in centimeters | From start of procedure through end of procedure (day 1)
Diagnostic yield of bronchoscopy utilizing a 3mm bronchoscope for eccentric lesions | Receipt of cytology/histopathology results (approximately 7 days)
  -Will be compared with historical controlled data of cases in which peripheral bronchoscopy was performed for peripheral lesions using radial probe EBUS and a 4mm bronchoscope in which eccentric ultrasound views were obtained
Ability to successfully convert ultrasound images from eccentric to concentric view by exchanging the 4mm thin bronchoscope for the 3mm ultrathin bronchoscope | From start of procedure through end of procedure (day 1)
  -The ability to convert will be based on the ultrasound image that is obtained using the 3mm bronchoscope (it will either be eccentric or concentric) compared to the eccentric ultrasound image obtained with the 4mm bronchoscope
Types of deficiencies associated with medical device | From start of procedure through end of procedure (day 1)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Chen, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu